CLINICAL TRIAL: NCT05143242
Title: A Randomized Controlled Trial Comparing Guided Bone Regeneration With Connective Tissue Graft to Re-establish Buccal Convexity at Implant Sites: Three-year Results.
Brief Title: Contour Augmentation by Means of Connective Tissue Grafting Versus Guided Bone Regeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-186
Record Dates: First submitted 2021-04-05; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Guided Bone Regeneration
Keywords: connective tissue graft; dental implant; guided bone regeneration; single tooth

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: Patients will be randomly assigned to the control group (GBR) or test group (CTG). Simple randomization was performed using sealed envelopes with an equal number of envelopes for every treatment group. Group allocation was revealed just prior to surgery by the surgeon.
  The measuring clinician will not be involved in the treatment of any of the patients and will be blinded to allow unbiased registrations.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided bone regeneration: Control (Active Comparator): Deproteinized bovine derived xenograft (Geistlich Bio-Oss® 0.25 - 1 mm, Geistlich Pharma AG, Wolhusen, Switzerland)
  Interventions: Procedure: Hard tissue augmentation at the buccal aspect of single implants.
- Connective tissue graft: Test (Active Comparator): Connective tissue graft harvested from the palate
  Interventions: Procedure: Soft tissue augmentation at the buccal aspect of single implants.

INTERVENTIONS:
Procedure: Hard tissue augmentation at the buccal aspect of single implants. — One or two releasing incisions are made. The periosteum is released and multiple bone perforations are made in the buccal bone prior to the application of deproteinized bovine derived xenograft. A Creos® membrane (Nobel Biocare, Gothenburg, Sweden) is used to cover the occlusal part of the alveolar crest and the xenograft particles. Finally, multiple single monofilament sutures are used for primary tension-free wound closure.
  Arms: Guided bone regeneration: Control
Procedure: Soft tissue augmentation at the buccal aspect of single implants. — A CTG is taken from the palate and transplanted to the buccal side between the alveolar bone and the buccal flap. The CTG is secured with single monofilament sutures.
  Arms: Connective tissue graft: Test

SUMMARY:
The most frequent aesthetic complication following single implant treatment seems to be a lack of buccal convexity. This 'alveolar process deficiency' is the result of buccal bone remodeling following tooth extraction.

A traditional approach to treat alveolar process deficiency is guided bone regeneration (GBR), however post-operative complications such as swelling, bleeding and pain are common and the aesthetic outcome may not be optimal.

An alternative to the traditional GBR approach could be soft tissue contour augmentation using a connective tissue graft (CTG) at the buccal aspect. Possible advantages over GBR include less morbidity at the implant site, a superior aesthetic outcome since there is no need for vertical releasing incisions and less costs since there are no biomaterials to be used.

The primary study objective is to compare the GBR and CTG group in terms of 2 and 3 dimensional tissue alterations, focusing on the amount of tissue gain and volume stability over time. The secondary study objectives are morbidity, overall radiographic, clinical and aesthetic outcomes.

DETAILED DESCRIPTION:
Aim:

This study aims to compare guided bone regeneration (GBR) with connective tissue graft (CTG) to re-establish buccal convexity at single implants.

Sample size calculation:

The sample size calculation was based on the primary study outcome (BSP) and was performed in SAS Power using the Satterthwaite t-test (De Bruyckere et al., 2018). The calculation was based on finding a mean difference of at least 0.5 mm between these groups with a standard deviation of 0.5 mm. This standard deviation was arbitrarily chosen given the lack of comparative studies. Alpha was set at 0.05 and the power was set at 0.80. This resulted in the inclusion of at least 17 patients per group. To compensate for possible drop-outs, 21 patients were included in each group.

Randomization and allocation concealment:

Patients were randomly assigned to the control group (GBR) or test group (CTG). Simple randomization was performed using sealed envelopes with an equal number of envelopes for every treatment group. Group allocation was revealed just prior to surgery by the surgeon and remained concealed for the evaluating investigator during the analytical stage of the project.

Surgical procedure:

In brief, a mucoperiosteal flap was raised in the control group by means of a midcrestal incision, sulcular incisions at both neighbouring teeth and a vertical parapapillary releasing incision at the distal neighbouring tooth. Following implant installation (NobelActive®, Nobel Biocare, Gothenburg, Sweden), the buccal concavity was augmented with deproteinized bovine bone mineral (DBBM) (Bio-Oss®; 0.25 - 1mm; Geistlich Biomaterials, Wolhusen, Switserland) and a collagen membrane (Creos® xenoprotect; 15x20mm; Nobel Biocare, Gothenburg, Sweden). Following apical release of the tissues, a cover screw was installed and primary wound closure was achieved (Seralon® 5/0, Serag Weissner, Naila, Germany). Aftercare included the use of a chlorhexidine rinse, systemic antibiotics (amoxicillin 1g, two times a day) and anti-inflammatory medication (ibuprofen 600mg) as deemed necessary by the patient. After 3 months, the implant was uncovered by means of a pouch procedure. A screw-retained provisional crown was placed as described by De Rouck et al. (2008), which was replaced by the permanent restoration (Procera® on ASC® abutment, Nobel Biocare, Gothenburg, Sweden) 3 months later.

The flap design in the test group was identical to the one in the control group, yet without a vertical parapapillary releasing incision. Instead of augmenting with DBBM, an appropriately sized CTG harvested from the palatal flap or palatal mucosa in the premolar area was pulled into the envelope and immobilized (Seralon® 5/0, Serag Weissner, Naila, Germany). Non-submerged healing was respected. Aftercare and prosthetic procedures were identical in both groups. All surgical treatments and provisional restorations were performed by the same clinician. Referring dentists made permanent restorations.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* Good oral hygiene defined as full-mouth plaque score ≤ 25% (O'Leary et al.1972
* Presence of a single tooth gap in the anterior maxilla (15 - 25) with both neighbouring teeth present
* Failing tooth at least 3 months earlier removed
* Class I defect at the single tooth gap as clinically assessed (buccopalatal loss of tissue with a normal apicocoronal ridge height) (Seibert, 1983)
* Signed informed consent
* Buccopalatal bone dimension of at least 6 mm at the central and crestal aspect of the single tooth gap to ensure complete embedding of an implant by bone

Exclusion Criteria:

* Systemic diseases
* Smoking
* (History of) periodontal disease
* Untreated caries lesions
* Need for horizontal bone augmentation at the time of implant placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Buccal soft tissue profile | Year 1 and 3
  The volumetric analysis software (Swissmeda/SMOP, Zürich, Switzerland) calculated a mean dimensional change (mm3) within the AOI (area of interest) for each patient at T5 (3 years). Given the variable size in AOI (mm2) among patients, the mean dimensional change per area was transformed to a mean linear change in buccal soft tissue profile (BSP) in mm.

SECONDARY OUTCOMES:
Midfacial recession | Month 6; Year 1 and 3
  Midfacial recession was registered between 6 months, 1 year and 3 years on the basis of digital surface models in STL format superimposed and imported in designated software (Swissmeda/SMOP, Zürich, Switzerland). Midfacial recession was calculated by subtracting the data from 1 and 3 years to 6 months of follow-up.
Buccal bone thickness | Year 1 and 3
  The thickness of the buccal bone was measured (in mm) at t2 (1 year) and t3 (3 years) perpendicular to the long axis of the implant. Buccal bone was measured from the implant surface to the bone-soft tissue interface at 3 levels.
Buccal soft tissue thickness | Year 1 and 3
  The thickness of the soft tissues was measured (in mm) at t2 (1 year) and t3 (3 years) perpendicular to the long axis of the implant. Buccal soft tissue thickness was measured from the bone-soft tissue interface to the buccal soft tissue outline at the same levels as buccal bone thickness.
Pink Esthetic Score | Year 1 and 3
  The PES awards 7 parameters: mesial papilla, distal papilla, soft tissue level, soft tissue contour, alveolar process deficiency, soft tissue colour, soft tissue texture. Each parameter is assessed with a 0-1-2 score, yielding a PES score ranging from 0 (worst aesthetic outcome) to 14 (perfect aesthetic outcome).
Mucosal Scarring Index | Year 1 and 3
  The MSI is a composite index based on five parameters: width, height/contour, colour, suture marks and overall appearance. Each parameter is assessed with a 0-1-2 score, yielding an MSI score ranging from 0 (no scar) to 10 (most extreme scar).
Marginal bone loss | Year 1 and 3
  Marginal bone loss was recorded at the mesial and distal aspect of each implant. The distance from the implant-abutment interface to the first bone-to-implant contact (so-called bone level) was assessed on peri-apical radiographs taken with the long-cone paralleling technique. Mesial and distal values were averaged to receive one value per implant.
Probing depth | Year 1 and 3
  Probing depth was registered at four locations (mesiobuccal, buccal, distobuccal and palatal) around the implant to the nearest 0.5 mm. A mean value was calculated per implant.
Plaque | Year 1 and 3
  Plaque was assessed at four locations (mesiobuccal, buccal, distobuccal and palatal) around the implant. Each location was scored 0 or 1 (the absence or presence of plaque, respectively). Plaque was expressed as a percentage.
Bleeding on probing | Year 1 and 3
  Bleeding on probing was assessed at four locations (mesiobuccal, buccal, distobuccal and palatal) around the implant. Each location was scored 0 or 1 (the absence or presence of bleeding, respectively). Bleeding on probing was expressed as a percentage.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akcali A, Schneider D, Unlu F, Bicakci N, Kose T, Hammerle CH. Soft tissue augmentation of ridge defects in the maxillary anterior area using two different methods: a randomized controlled clinical trial. Clin Oral Implants Res. 2015 Jun;26(6):688-95. doi: 10.1111/clr.12368. Epub 2014 Apr 10. PMID 24720375
- [Background] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354
- [Background] Buser D, Weber HP, Lang NP. Tissue integration of non-submerged implants. 1-year results of a prospective study with 100 ITI hollow-cylinder and hollow-screw implants. Clin Oral Implants Res. 1990 Dec;1(1):33-40. doi: 10.1034/j.1600-0501.1990.010105.x. PMID 2099210
- [Background] Buser D, Chappuis V, Kuchler U, Bornstein MM, Wittneben JG, Buser R, Cavusoglu Y, Belser UC. Long-term stability of early implant placement with contour augmentation. J Dent Res. 2013 Dec;92(12 Suppl):176S-82S. doi: 10.1177/0022034513504949. Epub 2013 Oct 24. PMID 24158332
- [Background] Buser D, Chappuis V, Bornstein MM, Wittneben JG, Frei M, Belser UC. Long-term stability of contour augmentation with early implant placement following single tooth extraction in the esthetic zone: a prospective, cross-sectional study in 41 patients with a 5- to 9-year follow-up. J Periodontol. 2013 Nov;84(11):1517-27. doi: 10.1902/jop.2013.120635. Epub 2013 Jan 24. PMID 23347346
- [Background] Chappuis V, Rahman L, Buser R, Janner SFM, Belser UC, Buser D. Effectiveness of Contour Augmentation with Guided Bone Regeneration: 10-Year Results. J Dent Res. 2018 Mar;97(3):266-274. doi: 10.1177/0022034517737755. Epub 2017 Oct 26. PMID 29073362
- [Background] Cosyn J, Eghbali A, De Bruyn H, Collys K, Cleymaet R, De Rouck T. Immediate single-tooth implants in the anterior maxilla: 3-year results of a case series on hard and soft tissue response and aesthetics. J Clin Periodontol. 2011 Aug;38(8):746-53. doi: 10.1111/j.1600-051X.2011.01748.x. PMID 21752044
- [Background] Cosyn J, Eghbali A, De Bruyn H, Dierens M, De Rouck T. Single implant treatment in healing versus healed sites of the anterior maxilla: an aesthetic evaluation. Clin Implant Dent Relat Res. 2012 Aug;14(4):517-26. doi: 10.1111/j.1708-8208.2010.00300.x. Epub 2010 Jul 17. PMID 20662859
- [Background] De Bruyckere T, Eghbali A, Younes F, De Bruyn H, Cosyn J. Horizontal stability of connective tissue grafts at the buccal aspect of single implants: a 1-year prospective case series. J Clin Periodontol. 2015 Sep;42(9):876-882. doi: 10.1111/jcpe.12448. Epub 2015 Sep 16. PMID 26373422
- [Background] De Bruyckere T, Eeckhout C, Eghbali A, Younes F, Vandekerckhove P, Cleymaet R, Cosyn J. A randomized controlled study comparing guided bone regeneration with connective tissue graft to re-establish convexity at the buccal aspect of single implants: A one-year CBCT analysis. J Clin Periodontol. 2018 Nov;45(11):1375-1387. doi: 10.1111/jcpe.13006. PMID 30133718
- [Background] De Bruyckere T, Cabeza RG, Eghbali A, Younes F, Cleymaet R, Cosyn J. A randomized controlled study comparing guided bone regeneration with connective tissue graft to reestablish buccal convexity at implant sites: A 1-year volumetric analysis. Clin Implant Dent Relat Res. 2020 Aug;22(4):468-476. doi: 10.1111/cid.12934. Epub 2020 Jul 19. PMID 32686234
- [Background] De Rouck T, Collys K, Cosyn J. Single-tooth replacement in the anterior maxilla by means of immediate implantation and provisionalization: a review. Int J Oral Maxillofac Implants. 2008 Sep-Oct;23(5):897-904. PMID 19014160
- [Background] Eghbali A, De Bruyn H, Cosyn J, Kerckaert I, Van Hoof T. Ultrasonic Assessment of Mucosal Thickness around Implants: Validity, Reproducibility, and Stability of Connective Tissue Grafts at the Buccal Aspect. Clin Implant Dent Relat Res. 2016 Feb;18(1):51-61. doi: 10.1111/cid.12245. Epub 2014 Jul 17. PMID 25040828
- [Background] Eghbali A, Seyssens L, De Bruyckere T, Younes F, Cleymaet R, Cosyn J. A 5-year prospective study on the clinical and aesthetic outcomes of alveolar ridge preservation and connective tissue graft at the buccal aspect of single implants. J Clin Periodontol. 2018 Dec;45(12):1475-1484. doi: 10.1111/jcpe.13018. Epub 2018 Nov 5. PMID 30290007
- [Background] Furhauser R, Florescu D, Benesch T, Haas R, Mailath G, Watzek G. Evaluation of soft tissue around single-tooth implant crowns: the pink esthetic score. Clin Oral Implants Res. 2005 Dec;16(6):639-44. doi: 10.1111/j.1600-0501.2005.01193.x. PMID 16307569
- [Background] Hammerle CH, Araujo MG, Simion M; Osteology Consensus Group 2011. Evidence-based knowledge on the biology and treatment of extraction sockets. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:80-2. doi: 10.1111/j.1600-0501.2011.02370.x. PMID 22211307
- [Background] Hanser T, Khoury F. Alveolar Ridge Contouring with Free Connective Tissue Graft at Implant Placement: A 5-Year Consecutive Clinical Study. Int J Periodontics Restorative Dent. 2016 Jul-Aug;36(4):465-73. doi: 10.11607/prd.2730. PMID 27333003
- [Background] O'Leary TJ, Drake RB, Naylor JE. The plaque control record. J Periodontol. 1972 Jan;43(1):38. doi: 10.1902/jop.1972.43.1.38. No abstract available. PMID 4500182
- [Background] Schneider D, Ender A, Truninger T, Leutert C, Sahrmann P, Roos M, Schmidlin P. Comparison between clinical and digital soft tissue measurements. J Esthet Restor Dent. 2014 May-Jun;26(3):191-9. doi: 10.1111/jerd.12084. Epub 2013 Dec 17. PMID 24341747
- [Background] Seibert JS. Reconstruction of deformed, partially edentulous ridges, using full thickness onlay grafts. Part I. Technique and wound healing. Compend Contin Educ Dent (Lawrenceville). 1983 Sep-Oct;4(5):437-53. No abstract available. PMID 6578906
- [Background] Thoma DS, Buranawat B, Hammerle CH, Held U, Jung RE. Efficacy of soft tissue augmentation around dental implants and in partially edentulous areas: a systematic review. J Clin Periodontol. 2014 Apr;41 Suppl 15:S77-91. doi: 10.1111/jcpe.12220. PMID 24641003
- [Background] Thoma DS, Naenni N, Benic GI, Hammerle CH, Jung RE. Soft tissue volume augmentation at dental implant sites using a volume stable three-dimensional collagen matrix - histological outcomes of a preclinical study. J Clin Periodontol. 2017 Feb;44(2):185-194. doi: 10.1111/jcpe.12635. Epub 2017 Jan 3. PMID 27716970
- [Background] Thoma DS, Bienz SP, Figuero E, Jung RE, Sanz-Martin I. Efficacy of lateral bone augmentation performed simultaneously with dental implant placement: A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:257-276. doi: 10.1111/jcpe.13050. PMID 30675733
- [Background] Tonetti MS, Cortellini P, Graziani F, Cairo F, Lang NP, Abundo R, Conforti GP, Marquardt S, Rasperini G, Silvestri M, Wallkamm B, Wetzel A. Immediate versus delayed implant placement after anterior single tooth extraction: the timing randomized controlled clinical trial. J Clin Periodontol. 2017 Feb;44(2):215-224. doi: 10.1111/jcpe.12666. Epub 2017 Jan 31. PMID 27978602
- [Background] Van der Weijden F, Dell'Acqua F, Slot DE. Alveolar bone dimensional changes of post-extraction sockets in humans: a systematic review. J Clin Periodontol. 2009 Dec;36(12):1048-58. doi: 10.1111/j.1600-051X.2009.01482.x. PMID 19929956
- [Background] Wessels R, De Roose S, De Bruyckere T, Eghbali A, Jacquet W, De Rouck T, Cosyn J. The Mucosal Scarring Index: reliability of a new composite index for assessing scarring following oral surgery. Clin Oral Investig. 2019 Mar;23(3):1209-1215. doi: 10.1007/s00784-018-2535-6. Epub 2018 Jul 3. PMID 29971512
- [Background] Wiesner G, Esposito M, Worthington H, Schlee M. Connective tissue grafts for thickening peri-implant tissues at implant placement. One-year results from an explanatory split-mouth randomised controlled clinical trial. Eur J Oral Implantol. 2010 Spring;3(1):27-35. PMID 20467596
- [Background] Zeltner M, Jung RE, Hammerle CH, Husler J, Thoma DS. Randomized controlled clinical study comparing a volume-stable collagen matrix to autogenous connective tissue grafts for soft tissue augmentation at implant sites: linear volumetric soft tissue changes up to 3 months. J Clin Periodontol. 2017 Apr;44(4):446-453. doi: 10.1111/jcpe.12697. Epub 2017 Feb 11. PMID 28107560